CLINICAL TRIAL: NCT05666245
Title: Evaluating Modes of Influenza Transmission Through the Conduct of Controlled Human Influenza Virus Infection Transmission Trials (CHIVITTs)
Brief Title: DMID 21-0041; Influenza CVD 59000
Acronym: EMIT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Wilbur Chen, MD, MS, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: HP-00103865; U19AI162130 (NIH)
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Personal Protective Equipment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Donors (Other): Donors are persons naturally infected with influenza.
  Interventions: Behavioral: No Intervention - Under High Air Hygiene; Behavioral: No Intervention - Under Low Air Hygiene
- Intervention Recipients (Experimental): Intervention recipients are participants who do not have influenza and will use personal protective equipment.
  Interventions: Behavioral: Personal Protective Equipment (PPE) - Under High Air Hygiene; Behavioral: Personal Protective Equipment (PPE) - Under Low Air Hygiene
- Control Recipients (No Intervention): Control recipients are participants who do not have influenza and will not be using personal protective equipment.

INTERVENTIONS:
Behavioral: Personal Protective Equipment (PPE) - Under High Air Hygiene — Intervention Recipients (IRs) will be required to wear a lightweight plastic face shield, comply with hand hygiene (i.e., using a hand sanitization product every 15 minutes, plus periodic hand washing with soap and water), and avoid face touching during each planned exposure event. The face shield may only be removed after leaving the exposure room to go to the bathroom, for other short comfort breaks, and at mealtimes. In these instances, hand hygiene will be used after removing or replacing the face shield; and Donors will not be present. Hand washing with soap and water will be required before meals. IR will be separated from Donors by more than 6 feet during meals. The exposure room will be supervised by a trained member of the study staff who will monitor to ensure that Intervention Recipients wear the face shield continuously, are separated from Donors at meals, and do not touch their faces.
  High air hygiene is achieved by filtration and/or use of germicidal UV-C.
  Arms: Intervention Recipients
Behavioral: No Intervention - Under High Air Hygiene — No intervention
  High air hygiene is achieved by filtration and/or use of germicidal UV-C.
  Arms: Donors
Behavioral: Personal Protective Equipment (PPE) - Under Low Air Hygiene — Intervention Recipients (IRs) will be required to wear a lightweight plastic face shield, comply with hand hygiene (i.e., using a hand sanitization product every 15 minutes, plus periodic hand washing with soap and water), and avoid face touching during each planned exposure event. The face shield may only be removed after leaving the exposure room to go to the bathroom, for other short comfort breaks, and at mealtimes. In these instances, hand hygiene will be used after removing or replacing the face shield; and Donors will not be present. Hand washing with soap and water will be required before meals. IR will be separated from Donors by more than 6 feet during meals. The exposure room will be supervised by a trained member of the study staff who will monitor to ensure that Intervention Recipients wear the face shield continuously, are separated from Donors at meals, and do not touch their faces.
  Low air hygiene is achieved with minimal ventilation.
  Arms: Intervention Recipients
Behavioral: No Intervention - Under Low Air Hygiene — No intervention
  Low air hygiene is achieved with minimal ventilation.
  Arms: Donors

SUMMARY:
The primary objective of EMIT-2 is to use a randomized controlled trial (RCT) design to implement interventions which are known to reduce inhalation (airborne) transmission, so that the contribution of transmission by route of aerosols for influenza may be identified.

ELIGIBILITY:
For Donors:

Inclusion Criteria:

* Provides written informed consent, able to comply with the planned study procedures, available for between 2 and 5 days stay in the research quarantine unit for the CHIVITT, and have the ability to attend the scheduled follow-up visits.
* Subjects must be able to comprehend the study requirements, as evidenced by a score of ≥70% or better on the comprehension assessment (two attempts permitted).
* Males and non-pregnant, non-breastfeeding females1 aged ≥18 and ≤59 years of age, at time of initial consent.

  *Pregnancy and breastfeeding status to be determined by self-report
* Laboratory-confirmed influenza infection within the past 48 hours at time of entry into the exposure event.

  *A rapid antigen test in the setting of known local influenza activity and with symptoms suggestive of influenza at that time is acceptable
* Within the past 48 hours at time of entry into the exposure event, onset of influenza-like illness, as defined as fever (measured oral temperature of ≥100.2°F or self-reported fever in the absence of a measured temperature) AND cough or sore throat, or onset of less specific symptoms with a positive molecular test for influenza virus infection
* No self-reported or known history of alcohol or drug abuse within the past two years and no illicit drug use within the last 30 days.
* Do not have clinically significant medical, psychiatric, and chronic or intermittent health conditions including those listed in Exclusion Criteria.
* Does not have an ongoing symptomatic condition for which subject has had or has ongoing medical investigations but has not yet received a diagnosis or treatment plan.

  *e.g., ongoing and debilitating fatigue without a diagnosis for the symptom.
* Agrees to the collection of specimens for secondary research.

Exclusion Criteria:

* Female of childbearing potential who is breastfeeding or has positive urine pregnancy test upon admission to the hotel quarantine unit.
* Presence of self-reported or medically documented significant medical or psychiatric condition(s)5

  *Significant medical or psychiatric conditions include but are not limited to:

  a. Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma, cystic fibrosis) requiring daily medications6 currently or any treatment of respiratory disease exacerbations or hospitalizations for acute respiratory illnesses (e.g., asthma exacerbation) in the last 5 years.
* Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short-acting beta agonists, theophylline, ipratropium, biologics.

  b. Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.

  c. Neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, seizures, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis).

  d. Ongoing malignancy or recent diagnosis of malignancy, including leukemia; treated, non-melanoma skin cancers are permissible.

  e. An autoimmune disease. f. An immunodeficiency of any cause. g. A blood disorder (e.g., sickle cell disease) h. Endocrine disorders (e.g., diabetes) i. Liver, kidney, metabolic disorders j. BMI ≥40 kg/m2 k. Any other condition or behavior that in the opinion of the PI would affect the ability to participate in the transmission study over the next several days.
* Presence of immunosuppression or any medications that may be associated with impaired immune responsiveness7.
* Including, but not limited to, corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids or other similar or toxic drugs during the preceding 12-month period. Low dose topical and intranasal steroid preparations used for a discrete period are permitted.
* Is a habitual smoker8 of tobacco, marijuana, or e-cigarettes per self-report.

  * Habitual smokers are those who smoke or vape more than four cigarettes, other tobacco products, e-cigarettes or marijuana in a week for more than three months or use an inhaled nicotine or marijuana product more than 3 days a week on average. Edible or patch forms of tobacco or marijuana products do not constitute an exclusion.
* Known allergy or intolerance to treatments for influenza and other respiratory infections (including but not limited to acetaminophen/paracetamol).
* History of a previous severe allergic reaction to medicines of any kind with generalized urticaria, angioedema, or anaphylaxis.
* Presence of co-infection with SARS-CoV-2, as detected via a multiplex nucleic acid amplification test (e.g., Biofire).
* Participating in any other interventional clinical research study that has a scheduled intervention 30 days prior to the CHIVITT or 30 after discharge from the research quarantine unit.
* Any condition, to include medical and psychiatric conditions, that in the opinion of the Investigator, might interfere with the safety of the subject or the study objectives.

For Recipients:

Inclusion Criteria:

* Enrolled in the Recipient Protocol (University of Maryland, Baltimore Institutional Review Board HP-97730)
* Provides written informed consent, able to comply with the planned study procedures, be available for an up to ~14-day stay for the CHIVITT and have the ability to attend the scheduled follow-up visits.
* Subjects must be able to comprehend the study requirements, as evidenced by a score of ≥70% or better on the comprehension assessment (two attempts permitted).
* No change in smoker status, alcoholism, or illicit drug use status, as compared from their responses collected during screening (EMIT-2 Recipient Protocol). (Prescribed stimulants for the treatment of attention deficit hyperactivity disorder [ADHD] and cannabinoids use do not constitute exclusionary criteria)
* No significant change (for the worse) in general health history or in concomitant medication use, as compared from their responses collected during screening (EMIT-2 Recipient Protocol).
* Agree not to meet with other participants (recipients or donors) outside of the programmed exposure events during the course of their participation in the CHIVITT.

Exclusion Criteria:

* Female of childbearing potential who has a positive urine pregnancy test within 24 hours of admission to the hotel quarantine unit or is breastfeeding or planning to become pregnant within 2 months after entry into a CHIVITT.
* Presence of infection with influenza, SARS-CoV-2, or other respiratory pathogens detected via a multiplex nucleic acid amplification test (e.g., Biofire) at admission to the hotel quarantine facility.
* Within the past 72 hours, presence of influenza-like illness, as defined as fever of ≥100.2°F AND cough or sore throat, in the absence of an alternative cause.
* Receipt of any blood products within the past 2 months.
* Does not agree to provide permission for secondary research use of extra samples collected and stored specimens.
* Habitual smoker of tobacco, marijuana, or e-cigarettes per self-report. (Habitual smokers are those who smoke or vape more than four cigarettes, other tobacco products, e-cigarettes or marijuana in a week for more than three months or use an inhaled nicotine or marijuana product more than 3 days a week on average. Edible or patch forms of tobacco or marijuana products do not constitute an exclusion.)
* Self-reported or known history of alcohol or drug abuse in the past two years and no illicit drug use within the last 30 days.
* Has an ongoing symptomatic condition1 for which the subject has had or has ongoing medical investigations but has not yet received a diagnosis or treatment plan.

  *e.g., ongoing chronic fatigue without a diagnosis for symptom.
* Presence of self-reported or medically documented significant medical or psychiatric condition(s)2

  *Significant medical or psychiatric conditions include but are not limited to:
  1. Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma, cystic fibrosis) requiring daily medications* currently or any treatment of respiratory disease exacerbations or hospitalizations for acute respiratory illnesses (e.g., asthma exacerbation) in the last 5 years.

     *Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short-acting beta agonists, theophylline, ipratropium, biologics.
  2. Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
  3. Neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, seizures, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis).
  4. Ongoing malignancy or recent diagnosis of malignancy, including leukemia; treated, non-melanoma skin cancers are permissible.
  5. An autoimmune disease.
  6. An immunodeficiency of any cause.
  7. A blood disorder (e.g., sickle cell disease)
  8. Endocrine disorders (e.g., diabetes)
  9. Liver, kidney, metabolic disorders
  10. BMI ≥40 kg/m2
  11. Any other condition or behavior that in the opinion of the PI would affect the ability to participate in the screening or future transmission studies.
* Presence of immunosuppression or any medications that may be associated with impaired immune responsiveness3.

  *Including, but not limited to, corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids or other similar or toxic drugs during the preceding 12-month period. Low dose topical and intranasal steroid preparations used for a discrete period are permitted.
* Known allergy or intolerance to treatments for influenza and other respiratory infections (including but not limited to oseltamivir, baloxavir, acetaminophen/paracetamol).
* History of a previous severe allergic reaction to medicines of any kind with generalized urticaria, angioedema, or anaphylaxis.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, University of Maryland School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - University of Maryland, College Park School of Public Health, College Park, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Donors | Control Recipients
Started | 6 | 28
Completed | 6 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donors | Control Recipients | Total
Number analyzed (Participants) | 6 | 28 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 28 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 1 | 17 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 10 | 13
  White | 2 | 14 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Nasal Swab [Count of Participants; unit: Participants] — Viral Testing for influenza infection was performed with molecular diagnostic testing of the nasal swab specimen; conducted on all Recipients to ascertain for transmission of influenza from Donors to Recipients. A total of 28 Recipients were evaluated with Viral Testing after exposure to a total of 6 Donors, who were confirmed to have influenza infection
  Participants | 6 | 28 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 4 | 26 | 30
  Unknown or Not Reported | 0 | 0 | 0
Influenza Symptoms Score [Count of Participants; unit: Participants] — Symptoms of influenza illness were collected from Recipients to ascertain for transmission of influenza infection from Donors to Recipients. The symptoms were collected with a twice daily completion of a Modified Jackson Score Investigator Assessment Tool and a once daily self-reported FLU-PRO Survey Instrument. A total of 28 Recipients were evaluated for Influenza Symptoms Score after exposure to a total of 6 Donors, who were confirmed to have influenza infection.
  Participants | 6 | 28 | 34
Serum HAI and FRNT antibody titers [Count of Participants; unit: Participants] — Serological evidence of influenza infection was performed from serum collected from Recipients for the measurement of hemagglutination inhibition (HAI) and focus reduction neutralization test (FRNT) antibody titers of Recipients to ascertain for transmission of influenza infection from Donors to Recipients. Serum was collected pre-exposure and post-exposure from a total of 28 Recipients to evaluate for serological evidence of influenza infection after exposure to a total of 6 Donors, who were confirmed to have influenza infection.
  Participants | 6 | 28 | 34

OUTCOME MEASURES:

1. Primary Outcome: Viral Confirmation
Description: Proportion of recipients with viral confirmation of influenza infection
Time Frame: 2 weeks
Population: A total of 28 Recipients (all under control conditions) were exposed to a total of 6 Donors.
Measure: Count of Participants; unit: Participants
Arm/Group | Donors | Control Recipients
Number analyzed (Participants) | 6 | 28
Participants | 6 | 0

2. Primary Outcome: Symptomatic Confirmation
Description: Proportion of recipients with symptomatic confirmation of influenza infection
Time Frame: 2 weeks
Population: A total of 28 Recipients (all under control conditions) were exposed to a total of 6 Donors.
Measure: Count of Participants; unit: Participants
Arm/Group | Donors | Control Recipients
Number analyzed (Participants) | 6 | 28
Participants | 6 | 0

3. Primary Outcome: Serological Confirmation
Description: Proportion of recipients with serological confirmation of influenza infection
Time Frame: 2 weeks
Population: A total of 28 Recipients (all under control conditions) were exposed to a total of 6 Donors.
Measure: Count of Participants; unit: Participants
Arm/Group | Donors | Control Recipients
Number analyzed (Participants) | 6 | 28
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, 12 weeks
Arm/Group | Donors | Control Recipients
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/28
Other Adverse Events (participants affected / at risk) | 1/6 | 10/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donors (N=6) | Control Recipients (N=28)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (3) — Elevated heart rate
Hypertension (Cardiac disorders) | 0 (0) | 7 (7) — Elevated blood pressure

LIMITATIONS AND CAVEATS:
The SARS-CoV-2 pandemic significantly interrupted seasonal influenza virus circulation during the years of the study, such that the hotel quarantine transmission study could only be conducted over 2 sequential influenza seasons (2022-23 and 2023-24). The 2022-23 season failed to identify a Donor due to the very early onset of local seasonal influenza that year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT05666245/Prot_000.pdf